CLINICAL TRIAL: NCT00074828
Title: A Comparison of the Oral Anticoagulant LY517717 Difumarate to Subcutaneous Enoxaparin for the Prevention of Venous Thromboembolic Events (VTE) Post-Total Hip Replacement (THR) and Post-Total Knee Replacement (TKR) Surgery
Brief Title: New Oral Anticoagulant Therapy for the Prevention of Blood Clots Following Hip or Knee Replacement Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8113; H8G-MC-EPBB
Record Dates: First submitted 2003-12-19; First posted 2003-12-23 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: Total Knee Replacement; Total Hip Replacement
Keywords: elective; primary unilateral
MeSH Terms: interventions — LY517717; Enoxaparin

ARMS (2):
- A (Experimental)
  Interventions: Drug: LY517717
- B (Active Comparator)
  Interventions: Drug: enoxaparin

INTERVENTIONS:
Drug: LY517717
  Arms: A
Drug: enoxaparin
  Arms: B

SUMMARY:
LY517717 (a capsule given by mouth) is a blood thinner that may prevent blood clots from forming in the legs and may prevent those blood clots from traveling to the lungs. Leg and lung blood clots occur commonly after patients have surgery to replace a hip or knee joint. These clots often occur while patients are in bed in the hospital after hip or knee joint surgery. The purpose of this study is to test if different dose strengths (amount of drug in the capsules) of LY517717 can prevent blood clots from forming and to determine if LY517717 is safe. This study will compare LY517717 to enoxaparin, another blood thinner. Enoxaparin is one of the standard medications given after hip or knee joint surgery.

ELIGIBILITY:
Inclusion Criteria:

* Are scheduled for total knee or hip replacement surgery (only one side, first time joint replacement)
* Are at least 18 years of age and no more than 75 years of age.
* Have a body weight more than 50 kg and less than 120 kg.
* Sign an approved Eli Lilly and Company informed consent document.

Exclusion Criteria:

* Have had hip or knee replacement surgery in the non-surgical leg or any surgical procedure in the surgical leg within 6 months prior to enrollment.
* Other surgeries (brain, spinal cord, eye within 12 months; chest or abdominal surgery within 1 month).
* Have taken drugs that might increase possibility of bleeding.
* Other risk factors for bleeding (bleeding disorders, abnormal results on blood tests, ulcers)
* Increased risk for blood clots.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2003-12; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of LY517717 to enoxaparin in the prevention of VTEs measured by the proportion of patients with VTE event (DVT and/or PE) as confirmed by bilateral venography or on clinical assessment | end of study drug administration

SECONDARY OUTCOMES:
Safety and tolerability, major and minor bleeding, death due to VTE, effect on QTc duration, AEs and SAEs, hepatobiliary and other safety lab parameters | baseline, daily during therapy, at follow up visit
Pharmacokinetics and pharmacodynamics | predose, daily during therapy
Compare the effect of LY517717 versus enoxaparin measured by DVT, Proximal DVT, Distal DVT and PE | end of study drug administration
Compare the effect of LY517717 versus enoxaparin with confirmed VTE | end of study drug administration
Compare the effect of LY517717 versus enoxaparin measured by all confirmed VTEs and /or clinically suspected and confirmed VTE | through follow up

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Nedlands, Western Australia, Australia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Vienna, Austria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Brussels, Belgium
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Ostrava-Poruba, Czechia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Aachen, Germany
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Kecskemét, Hungary
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Perugia, Italy
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Bydgoszcz, Poland

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com